CLINICAL TRIAL: NCT04627207
Title: A Randomized, Open, Single-dose, 3 Period Partial Replicated Crossover-design Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics After Administration of CKD-333 or Co-administration of CKD-330 and D085 in Healthy Volunteers Under Fasting Conditions
Brief Title: A Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics of CKD-333 or Co-administration of CKD-333 and D085 in Healthy Volunteers
Acronym: CKD-333
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A70_10BE2006
Record Dates: First submitted 2020-11-11; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Diseases
Keywords: CKD-333
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reference-Reference-Test (Experimental): Sequence 1
  Interventions: Drug: CKD-330 1 Tab. and D085 1 Tab.; Drug: CKD-333 1 Tab
- Reference-Test-Reference (Experimental): Sequence 2
  Interventions: Drug: CKD-330 1 Tab. and D085 1 Tab.; Drug: CKD-333 1 Tab
- Test-Reference-Reference (Experimental): Sequence 3
  Interventions: Drug: CKD-330 1 Tab. and D085 1 Tab.; Drug: CKD-333 1 Tab

INTERVENTIONS:
Drug: CKD-330 1 Tab. and D085 1 Tab. — Other names: Reference
Drug: CKD-333 1 Tab — Other names: Test

SUMMARY:
A clinical trial to evaluate the safety and pharmacokinetic characteristics of CKD-333 or Co-administration of CKD-333 and D085 in healthy volunteers

DETAILED DESCRIPTION:
A randomized, open, single-dose, 3 period partial replicated crossover-design clinical trial to evaluate the safety and pharmacokinetic characteristics after administration of CKD-333 or co-administration of CKD-330 and D085 in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19≤ ~ <55-year-old.
* Those who have body weight ≥ 55kg (men) or ≥ 45kg (women), with calculated body mass index(BMI) of 17.5 ≤ ~ < 30.5 kg/m2
* Those who have no congenital/chronic diseases, abnormal symptoms.
* Those who were deemed to eligible for participation of clinical trial by laboratory tests, vital signs and 12-lead ECG etc.
* Those who voluntarily decide to participate and agree to comply with the cautions and fully understanding the detailed description of this clinical trial.
* Those who consent to proper contraception during the study period and do not donate sperm until 14 days after the last administration of investigational product. And those who consent not to become pregnant or breastfeeding.
* Those who have ability and willingness to participate in clinical trial

Exclusion Criteria:

* Those who have medical history or medical symptom of liver, kidney, nervous system, respiratory system, digestive system, endocrine system, blood/tumor, urinary system, cardiovascular system, musculoskeletal disease, or mental disease.
* Those who have past medical history of gastrointestinal disorder (Crohn's disease, ulcerative colitis, etc. except simple appendectomy or hernia surgery), which affect the absorption of drug.
* Those who have the test results written below,

  * AST or ALT are 2 times higher than upper normal range
  * Creatinine is upper normal range or eGFR (estimated Glomerular Filtration Rate, which is calculated by MDRD) < 60 mL/min/1.73m2
  * QTc is higher than 450msec measured by 12-lead ECG
  * CPK is 3 times higher than upper normal range
  * Serum Potassium is higher than 5.5 mEq/L
  * Hematocrit is under normal range
* Those who exceed alcohol consumption criteria (21 units/week within 3 months) prior to first administration of investigational product. Or Those who can't quit drinking alcohol from 48 hours to end of bleeding time point.
* Those who exceed smoke criteria (20 cigarettes/day within 6 months) prior to first administration of investigational product. Or Those who can't quit smoking during hospitalization.
* Those who have participated in other clinical trial and received Investigational product within 6 month prior to the first administration of drug.
* Those who have the test results written below,

  * Systolic blood pressure ≥140 mmHg or <90 mmHg
  * Diastolic blood pressure ≥90 mmHg or <60 mmHg
* Those who have a drug abuse history within one year prior to first administration of investigational product or positive reaction on urine drug screening test.
* Those who take barbiturate and related (causing induction or inhibition of metabolism) drug within 1 month before the first administration of investigational product.
* Those who received following drugs, which may affect results of clinical trial and safety.

  * Ethical-the-counter (ETC) drugs or Over-the-counter (OTC) drugs within 10 days before the first administration of the investigational drug (especially Glecaprevir, Pibrentasvir).
* Those who donated whole blood within 2 months or apheresis within 1 month or received transfusion within 1 month.
* Those who have history of hypersensitivity to active pharmaceutical ingredient or Dihydropyridine or Aspirin, antibiotics etc.
* Those who deemed to ineligible for participation of clinical trial,

  * Patient with hyperkalemia
  * Patients with hepatopathy
  * Patients with hereditary angioedema, ACE inhibitors or angiotensin II receptor antagonists who have a history of angioedema
  * Primary hyperaldosteronism
  * Patients with aortic valve stenosis, mitral (valve) stenosis, hypertrophic obstructive cardiomyopathy
  * Patients with ischemic heart disease, ischemic cardiovascular disease, cerebrovascular disease
  * Patients with Intravascular volume depletion
  * Patients with diabetes or kidney failure
  * Patients with renal artery stenosis
  * Patients with muscle disease
  * Patients with Hypothyroidism
  * Patients with a history of muscle toxicity when using statins or fibrates
  * Patients who have recently had a kidney transplant
  * Patients with history of shock
* Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
* Those who took caffeine or grapefruit within 3 months(5 cups/day) (before the first administration of investigational product) and can't stop taking caffeine or grapefruit until the end of clinical trial.
* Those who can't eat standard meal during hospitalization.
* Those who are pregnant or breastfeeding.
* Those who are deemed to ineligible for participation of clinical trial by investigators.

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
AUCt of CKD-330, D085, CKD-333 | Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Area under the CKD-330/D085/CKD-333 concentration in blood-time curve from zero to final
Cmax of CKD-330, D085, CKD-333 | Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  The maximum CKD-330/D085/CKD-333 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jang Hee, M.D., Principal Investigator — Chungnam National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JH, Song JH, Kim M, Hong JH, Sunwoo J, Jung JG. Pharmacokinetic Comparison of a Fixed-Dose Combination of Candesartan Cilexetil/Amlodipine/Atorvastatin Versus Co-administration of Individual Formulations in Healthy Participants. Adv Ther. 2024 Jul;41(7):2808-2825. doi: 10.1007/s12325-024-02869-y. Epub 2024 May 21. PMID 38771476